CLINICAL TRIAL: NCT04851223
Title: Biomarkers Identification for the Progression From Pre-diabetes to T2D
Brief Title: Investigating Plasma Biomarker Molecules Associated With the Progression of Prediabetes to Overt Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roehampton (Other)
Responsible Party: Principal Investigator, Richard Mackenzie, Dr., University of Roehampton
Other Study IDs: LSC 20/ 311; 245301 (Other: IRAS ID)
Record Dates: First submitted 2021-01-14; First posted 2021-04-20 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Type2 Diabetes Mellitus; Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre Diabetics

SUMMARY:
There are an estimate 7 million people in the United Kingdom living with pre-diabetes. The increasing number of new cases of pre-diabetes presents a global health concern due to funding implications.

The progression from pre-diabetes to overt type 2 diabetes is often characterised by a reduction in insulin secretion (or β-cell dysfunction). Whilst inflammation may contribute to β-cell dysfunction, a complete picture is still lacking. The proposed research will help develop a more complete understanding of the molecules that may trigger β-cell failure, a process that often connects pre-diabetes to overt diabetes.

The aims of this project are;

1. Run large-scale proteomics and metabolomics analysis in pre-diabetic individuals to determine possible biomarker molecules.
2. Use measures and / or classifications of insulin resistance and diabetes (i.e. β-cell function and Disposition Index) to establish whether particular metabolic and / or proteomic signatures (aim 1) are associated with the development of pre-diabetes.
3. To determine if the possible metabolite or protein profile changes are associated with the progression or regression of pre-diabetes from baseline (0 month) to the end of the National Diabetes Prevention Programme (NDPP) (9 month).

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a complex metabolic disease characterised by elevated blood sugar. This represents a worldwide concern due to the secondary complications associated with type 2 diabetes, which are considered an important cause of early death; particularly, given the predicted increase. The cost associated with the treatment and the complications associated with diabetes reaches £10 billion every year and it is expected to increase. From approximately 425 million (2017) it is projected that 629 million adults will be living with diabetes by 2045. Therefore, this matter requires effective interventions aimed at improving blood sugar control, reducing the burden on the economy while improving the quality of life among T2DMs.

Insulin, a hormone that is allowing the body to use or store sugar derived from food, is manufactured by the β-cells in the pancreas. The progression from pre-diabetes to overt type 2 diabetes is typically diagnosed at the point of β-cell failure. Several factors are known to contribute to β-cell dysfunction such as: obesity (especially abdominal obesity), high blood pressure and elevated fats in the blood. Around 80% of the people who have been diagnosed with T2DM are either obese or overweight and they have been observed to have increased levels of fatty acids in the blood following a meal, which can induce insulin resistance. High levels of fatty acids have also been associated with an increased production of pro-inflammatory cytokines, which are small proteins that have an effect on organs or other cells, contributing to chronic inflammation. High levels of chronic inflammation increase the chances of developing metabolic disorders such as T2DM. However, a complete picture of this process is still lacking.

The proposed study will help develop a more complete understanding of the molecules that may trigger β-cell failure.

The identification of these molecules that are implicated in β-cell failure, can lead to the development of targeted interventions for those at risk of developing type 2 diabetes and potentially preventing habitual hyperglycaemia and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Pre-diabetic individuals between 18 and 65 years of age

Pre-diabetes criteria:

* Glycated hemoglobin (HbA1c) values between 42 - 47 mmol/mol
* Fasting plasma glucose levels between 6.1 - 6.9 mmol/L
* Blood pressure <140 mmHg systolic/ <90 mmHg diastolic

Exclusion Criteria:

* Individuals suffering from any complications (i.e. nerve or kidney disorders, damage of the retina, vascular diseases, strokes, persistent high blood pressure, cardiovascular disease,haemophilia), those with anaemia, blood borne diseases, those who are pregnant or in the postpartum period (within 3 months after delivery), have high blood pressure >140 mmHg systolic/ >90 mmHg diastolic, current smokers, individuals requiring strong anticoagulant medication, such as warfarin (the anticoagulant effect of non-steroidal anti-inflammatory drugs is too small to pose a hazard), insulin or other medications affecting the typical levels of blood glucose are unfortunately unable to take part in this study. Individuals must not be involved in any other study which involves the sampling of blood and must not have donated blood in the last 12 weeks (for males) or 16 weeks (for females). A health questionnaire will be carried out to confirm your eligibility for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-diabetic individuals
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-06-22 (Estimated); Study Completion 2023-09-22 (Estimated)

PRIMARY OUTCOMES:
Body weight Measurements | Changes from baseline to 6 and 9 months
  Weight in kilograms
Body mass Index measurements | Changes from baseline to 6 and 9 months
  kg/m^2
Changes in insulin and glucose | Changes from baseline to 6 and 9 months
  Effect of insulin and glucose levels expressed in mg/dl
Changes in BCAA and its derivatives | Changes from baseline to 6 and 9 months
  metabolites levels via mass spectrometry analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Roehampton, London, United Kingdom

REFERENCES:
- [Background] Mokdad AH, Ford ES, Bowman BA, Dietz WH, Vinicor F, Bales VS, Marks JS. Prevalence of obesity, diabetes, and obesity-related health risk factors, 2001. JAMA. 2003 Jan 1;289(1):76-9. doi: 10.1001/jama.289.1.76. PMID 12503980
- [Background] Reaven GM, Hollenbeck C, Jeng CY, Wu MS, Chen YD. Measurement of plasma glucose, free fatty acid, lactate, and insulin for 24 h in patients with NIDDM. Diabetes. 1988 Aug;37(8):1020-4. doi: 10.2337/diab.37.8.1020. PMID 3292322